CLINICAL TRIAL: NCT04957082
Title: Culturally-targeted Communication to Promote SARS-CoV-2 Antibody Testing in Saliva: Enabling Evaluation of Inflammatory Pathways in COVID-19 Racial Disparities
Brief Title: Culturally-Targeted COVID-19 Communication and SARS-CoV-2 Antibody Testing Evaluation and Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Todd Lucas, Principal Investigator, Michigan State University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: MSUSeronet1; U01CA260469 (NIH)
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: SARS-CoV2 Infection
Keywords: SARS-CoV-2; COVID-19; Health Disparities; Health Communication; Antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Design is partial factorial. All white participants and half of African American participants will receive general video education/messaging. Half of African American participants will be assigned to an intervention condition that includes culturally-targeted information about SARS-CoV-2 antibody testing.
Who Masked: Participant
Masking Description: Participants will be unaware of their assignment to a general versus culturally targeted condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White Flint Registry: General (Active Comparator): White participants receive "general consumption" video information about SARS-CoV-2 antibody testing.
  Interventions: Behavioral: General SARS-CoV-2 Communication
- African American Registry: General (Active Comparator): African American participants receive "general consumption" video information about SARS-CoV-2 antibody testing.
  Interventions: Behavioral: General SARS-CoV-2 Communication
- African American Registry: Culturally Targeted (Experimental): African American participants receive culturally targeted video information about SARS-CoV-2 antibody testing.
  Interventions: Behavioral: Culturally Targeted SARS-CoV-2 Communication

INTERVENTIONS:
Behavioral: Culturally Targeted SARS-CoV-2 Communication — SARS-CoV-2 video tutorial includes a one minute video based messaging adjunct meant to enact a culturally targeted framing of health information presented to African Americans.
  Arms: African American Registry: Culturally Targeted
Behavioral: General SARS-CoV-2 Communication — SARS-CoV-2 video tutorial is for general consumption and does not include culturally targeted information
  Arms: African American Registry: General; White Flint Registry: General

SUMMARY:
This disparities-focused study seeks to evaluate communication strategies for better encouraging understanding and uptake of salivary SARS-CoV-2 antibody testing among African Americans residing in Flint, Michigan. This iteration will consider individuals recruited from the Flint Registry and assess willingness to participate in a drive-up saliva sample collection taking place at a central location in Flint, Michigan.

DETAILED DESCRIPTION:
African Americans develop and die from SARS-CoV-2 infection more than any other racial group in the United States, including in majority African American cities such as Flint, Michigan. Addressing these disparities may be aided by SARS-CoV-2 antibody testing. However, African Americans may be reluctant to partake in conventional antibody testing programs due to medical mistrust and experiences with racism. This study seeks to evaluate communication strategies for better encouraging understanding and uptake of salivary SARS-CoV-2 antibody testing. The central hypothesis is that African-Americans will be more receptive to antibody testing when benefits and limitations are communicated in a culturally effective manner. Our clinical trial aims are to 1) develop and compare effects of a general versus culturally-targeted video about antibody testing on African American and White Flint residents' antibody testing attitudes and uptake; 2) identify and compare effects of a general versus culturally-targeted video on activation of medical mistrust and racism-related cognition among African Americans when considering antibody testing. In collaboration with clinical and community partners, we have prepared and will evaluate general and culturally-targeted video tutorials about SARS-CoV-2 antibody testing. These brief videos will be distributed to the Flint community through the Flint Registry - a highly visible local health resource exchange. We will furnish an opportunity to engage salivary antibody screening and measure willingness to participate. In this study iteration, we will consider willingness to participate in a drive-up saliva sample collection that is taking place at a central location in Flint, Michigan.

ELIGIBILITY:
Inclusion Criteria:

* African American or White, 18 or older, and enrolled in the Flint Registry

Exclusion Criteria:

* All who do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Flint Journal Building, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per requirements and sharing structures established by NCI "SeroNet" initiative.
Supporting Information: Analytic Code
Time Frame: Upon Study Completion

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
Started | 229 | 207 | 230
Completed | 198 | 128 | 161
Not Completed | 31 | 79 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted | Total
Number analyzed (Participants) | 198 | 128 | 161 | 487
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 168 | 113 | 142 | 423
  >=65 years | 30 | 15 | 19 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 73 | 104 | 277
  Male | 98 | 55 | 57 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 1 | 10
  Not Hispanic or Latino | 190 | 125 | 159 | 474
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 128 | 161 | 289
  White | 198 | 0 | 0 | 198
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number (Percentage) of Participants Requested to Participate in Saliva-based SARS-CoV-2 Antibody Testing
Description: Number (Percentage) of participants who respond "yes" to be included in offer to participate in no cost SAR-CoV-2 salivary antibody test.
Time Frame: Immediately following didactic study portion and health communication randomization on day 1.
Population: Number (percentage) of participants in each condition who opted to participate in salivary antibody testing.
Measure: Count of Participants; unit: Participants
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
Number analyzed (Participants) | 198 | 128 | 161
Participants | 175 | 84 | 121

2. Primary Outcome: Number (Percentage) of Participants Who Requested Saliva-based SARS-CoV-2 Antibody Testing Participated in the Testing.
Description: Number (Percentage) of participants that requested to participate in antibody testing who actually complete antibody testing.
Time Frame: 8 weeks from the day of consenting to participate in the salivary-based SARS-CoV-2 antibody testing
Measure: Count of Participants; unit: Participants
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
Number analyzed (Participants) | 175 | 84 | 121
Participants | 111 | 55 | 79

3. Primary Outcome: SARS-CoV-2 Antibody Testing Attitudes
Description: Submeasure of Theory of Planned Behavior Indicating extent of a favorable attitude SARS-CoV-2 towards antibody testing (Seven point Likert Rating, with higher scores indicating more favorable Attitudes).
Time Frame: Immediately following didactic study portion and health communication randomization on day 1.
Population: All participants for whom Theory of Planned Behavior measure was successfully recorded immediately following messaging randomization.
Measure: Mean (Standard Deviation); unit: Units on a Scale (Minimum:1, Maximum:7)
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
Number analyzed (Participants) | 198 | 128 | 161
Units on a Scale (Minimum:1, Maximum:7) | 5.91 (1.13) | 5.61 (1.31) | 5.71 (1.22)

4. Primary Outcome: SARS-CoV-2 Antibody Testing Normative Beliefs
Description: Sub-measure of Theory of Planned Behavior Indicating extent to which believes other people are favorable towards SARS-CoV-2 towards antibody testing (Seven point Likert Rating, with higher scores indicating stronger Normative Beliefs).
Time Frame: Immediately following didactic study portion and health communication randomization on day 1.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale (Minimum:1, Maximum:7)
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
Number analyzed (Participants) | 198 | 128 | 161
Units on a Scale (Minimum:1, Maximum:7) | 4.71 (1.38) | 4.69 (1.41) | 4.85 (1.45)

5. Primary Outcome: Antibody Testing Perceived Behavioral Control
Description: Sub-measure of Theory of Planned Behavior Indicating Self Efficacy to Complete Antibody Testing (Seven point Likert Rating, with higher scores indicating greater Perceived Behavioral Control).
Time Frame: Immediately following didactic study portion and health communication randomization on day 1.
Measure: Mean (Standard Deviation); unit: Units on a Scale (Minimum:1, Maximum:7)
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
Number analyzed (Participants) | 198 | 128 | 161
Units on a Scale (Minimum:1, Maximum:7) | 5.88 (1.19) | 5.71 (1.29) | 5.76 (1.37)

6. Primary Outcome: Antibody Testing Intentions
Description: Sub-measure of Theory of Planned Behavior indicating Intentions to Complete Antibody Testing (Seven point Likert Rating, with higher scores indicating stronger screening Intentions).
Time Frame: Immediately following didactic study portion and health communication randomization on day 1.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale (Minimum:1, Maximum:7)
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
Number analyzed (Participants) | 198 | 128 | 161
Units on a Scale (Minimum:1, Maximum:7) | 4.81 (1.52) | 4.61 (1.54) | 4.83 (1.57)

7. Primary Outcome: Antibody Testing Anticipatory Racism
Description: Extent to which participants believe that racism-related factors would diminish the value of SARS-CoV-2 antibody testing for self (Seven-point Likert rating, with higher scores indicating greater Anticipatory Racism).
Time Frame: Immediately following didactic study portion and health communication randomization on day 1.
Population: All participants for whom Anticipatory Racism measure was successfully recorded immediately following messaging randomization.
Measure: Mean (Standard Deviation); unit: Units on a Scale (Minimum:1, Maximum:7)
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
Number analyzed (Participants) | 198 | 128 | 161
Units on a Scale (Minimum:1, Maximum:7) | 1.79 (1.25) | 2.93 (1.54) | 2.94 (1.57)

ADVERSE EVENTS:
Time Frame: 8 weeks.
Arm/Group | White Flint Registry: General | African American Registry: General | African American Registry: Culturally Targeted
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/128 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/198 | 0/128 | 0/161
Other Adverse Events (participants affected / at risk) | 0/198 | 0/128 | 0/161

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT04957082/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT04957082/SAP_001.pdf